CLINICAL TRIAL: NCT03186547
Title: Satisfaction Of Adult Patients With Gummy Smile Treated By Botulinum Toxin A Injection Versus Modified Lip Repositioning Surgery : A Randomized Clinical Trial
Brief Title: Satisfaction Of Adult Patients With Gummy Smile Treated By Botulinum Toxin A Injection
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zeinab mohamed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-06-02
Record Dates: First submitted 2017-06-11; First posted 2017-06-14 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Gummy Smile Due to Hypermobile Upper Lip
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Botulinum Toxin A Injection (Experimental): this group will receive Botulinum Toxin A Injection at doses of 2.5 or 5 IU (depending on the degree of gum exposure) on each side of the nasolabial fold with follow up at at 2,4,8,12 and 24 weeks.
  Interventions: Drug: Botulinum Toxin A Injection
- Modified Lip Repositioning Surgery (Experimental): this group will receive Modified Lip Repositioning Surgery with follow up at at 2,4,8,12 and 24 weeks.
  Interventions: Procedure: Modified Lip Repositioning Surgery

INTERVENTIONS:
Drug: Botulinum Toxin A Injection — adult patients with gummy smile due to hypermobile upper lip will receive Botulinum Toxin A Injection with a single injection1 cm lateral to the ala horizontally and 3 cm above the lip line vertically.
  Other Names: BOTOX
  Arms: Botulinum Toxin A Injection
Procedure: Modified Lip Repositioning Surgery — the surgical procedure will be done by removal of strip of epithelium by careful dissection and stabilizing the new mucosal margin to the gingiva to improve the gingival display in adult patients with gummy smile.
  Arms: Modified Lip Repositioning Surgery

SUMMARY:
The aim of the proposal study is to answer the question of how to manage gummy smiles due to hypermobile upper lip with less invasive and low risk level procedure . This trial will help the practitioners and the patients in taking the convenient decision to correct the gumminess to restore lip-gingival-dental harmony and enhance smile asthetics.

DETAILED DESCRIPTION:
In this randomized clinical trial , two groups will be included to compare the effectiveness of a treatment modality of botulinum toxin-A injection , in the first group , on gingival display during smiling ,patient satisfaction , lower face esthetics ( upper lip length , upper lip vermillion length , interlabial gap , nasolabial angle) and the postoperative side effects . the comparator group will receive treatment by modified lip repositioning surgery ,to compare the results of the intervention group that can possibly obtained without undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults with age range from 18 - 30 years.
* Excessive gingival display more than 3 mm during smiling.
* Patients having hypermobile upper lip with or without (mild / moderate) vertical maxillary excess.
* Patients with normal morphology of clinical crowns.
* Normal lip separation (ILG) at rest
* Medically free subjects.

Exclusion Criteria:

* Patients with systemic diseases or neuromuscular disorders.
* Gummy smile with gingival display more than 8 mm during smiling.
* Severly long face (VME) patients.
* Patients with periodontal disease or gingival hyperplasia .
* Medically compromised patients contraindicated for surgery .
* Pregnant or lactating female patients.
* Patients with inadequate attached gingiva .

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction and postoperative side effects | at 4 weeks
  it will be assessed using Questionnaire.

SECONDARY OUTCOMES:
Improvement of gingival display upon smiling | at 4,8 and 12 weeks
  it will be assessed using Digital ruler on DSS software
Lower face esthatics: a) upper lip length b) upper lip- vermillion length c) interlabial gap | at 4,8 and 12 weeks
  it will be assessed using Digital ruler and angle measurement on DSS software
Lower face esthatics: d)nasolabial angle | at 4,8 and 12 weeks
  it will be assessed using Digital angle measurement on DSS software
stability of gummy smile correction. | at the end of 24 weeks.
  it will be assessed using Digital ruler on DSS software

IPD SHARING:
Plan to Share IPD: Yes